CLINICAL TRIAL: NCT02308930
Title: Effect of Dietary DHA Supplementation on Cognitive Performance and Growth in Chinese School Children: A Randomized Controlled Study
Brief Title: Effect of DHA Supplementation on Cognitive Performance and Growth in Chinese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huilian Zhu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TY0131002
Record Dates: First submitted 2014-11-30; First posted 2014-12-05 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Vitamins; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Vitamins + DHA supplement (Experimental): 2 x 400 mg capsules per day orally for 6 months, each capsule providing 154μg Vitamin A, 2.36μg Vitamin D, 0.4mg Vitamin E and 375mg algal oil (containing 150mg DHA).
  Interventions: Dietary Supplement: Vitamins + DHA supplement (Vitamins A,D, E and algal oil)
- Vitamins supplement (Other): 2 x 400 mg capsules per day orally for 6 months, each capsule providing 154μg Vitamin A, 2.36μg Vitamin D, 0.4mg Vitamin E and 375mg corn oil (free of omega-3 fatty acids).
  Interventions: Dietary Supplement: Vitamins supplement (Vitamins A,D, E and corn oil)

INTERVENTIONS:
Dietary Supplement: Vitamins + DHA supplement (Vitamins A,D, E and algal oil)
  Arms: Vitamins + DHA supplement
Dietary Supplement: Vitamins supplement (Vitamins A,D, E and corn oil)
  Arms: Vitamins supplement

SUMMARY:
The purpose of this study is to determine whether DHA supplement (in a daily dose of 300 mg) will improve the cognitive performance, associated metabolism and growth in normal children aged 6-12 years in primary schools.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-12 years from primary schools.
2. Healthy as assessed by a physician.
3. Willing to participate in the study, consume the test product and perform all measurements including cognitive testing, blood drawing, urine samples, anthropometry and questionnaires.
4. Willing to maintain current dietary habits and intend to stay in the study area for ≥ one year.
5. Informed consent signed by parent or caregiver and oral consent given by child.

Exclusion Criteria:

1. Children with obvious mental and physical handicaps.
2. Children taking medication which interferes with study measurements (e.g., psychoactive medications or medications expected to affect behavior and learning).
3. Taking dietary supplements already.
4. Suffering major life events (immediate family death, parents divorce, etc.) within six months.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Performance on Wisconsin card sorting test (WCST) and digit span test | 6 months
  At baseline, 3 and 6 months cognitive tests will be administered, and the scores of Wisconsin card sorting test (WCST) and digit span test will be recorded.

SECONDARY OUTCOMES:
DHA related metabolites and neurotransmitters (blood concentration of DHA related metabolites and neurotransmitters) | 6 months
  At baseline and 6 months, blood samples will be drawn and the concentration of DHA related metabolites and neurotransmitters will be detected using biochemical methods.

REFERENCES:
- [Derived] Yang GY, Wu T, Huang SY, Huang BX, Wang HL, Lan QY, Li CL, Zhu HL, Fang AP. No effect of 6-month supplementation with 300 mg/d docosahexaenoic acid on executive functions among healthy school-aged children: a randomized, double-blind, placebo-controlled trial. Eur J Nutr. 2021 Jun;60(4):1985-1997. doi: 10.1007/s00394-020-02388-w. Epub 2020 Sep 26. PMID 32979077